CLINICAL TRIAL: NCT07046793
Title: Fracture Ultrasound in Kids Wirst Trial (FRUSKI-Wrist)
Acronym: FRUSKI-Wrist
Status: Completed | Type: Observational
Sponsor: David Troxler (Other)
Collaborators: Luzerner Kantonsspital (Other); Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Geneva (Other); La Tour Hospital (Other); Hôpital Fribourgeois (Other); University Children's Hospital Basel (Other)
Responsible Party: Sponsor-Investigator, David Troxler, Sponsor Investigator, University Children's Hospital Basel
Organization: University Children's Hospital Basel (Other)
Other Study IDs: 2022-00376
Record Dates: First submitted 2025-06-29; First posted 2025-07-02 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Fractures in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: POCUS — Ultrasound screening of the distal forearm.

SUMMARY:
This is a multicenter combined diagnostic accuracy study and observational prospective cohort.

Part one aims to confirm non-inferiority of POCUS for the detection of distal forearm fractures compared to X-ray.

Part two aims to confirm non-inforiority of POCUS compared to x-ray for the detection of potentially unstable forearm fractures needing follow up imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency room of a study hospital with an acute trauma to the wrist and suspected fracture of the wrist consulted by a trained study examiner.
* Age 0-18 years Depending on the result

Exclusion Criteria:

* Patient needing immediate medical attention (triage score 1 or 2) as well as severely displaced or open fractures or neurovascular compromise distally to the suspected fracture.
* Patient with imaging studies obtained prior to the emergency room visit
* Patient with prior fracture of the affected wrist within the last 24 months
* Patient refusing participation / missing informed consent.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with wrist trauma
Sampling Method: Non-Probability Sample
Enrollment: 815 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Fracture yes/no as final diagnosis | at 4 weeks from inclusion
Possible unstable fracture as final diagnosis | 4 weeks from inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Kinderspital zentralschweiz, Lucerne, Switzerland